CLINICAL TRIAL: NCT07008664
Title: Signature Development and Validation Protocol for an Epigenetic Assay in Diagnosing Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: EPOCH Epigenetics, Inc (Unknown)
Responsible Party: Principal Investigator, Jeffrey Marshall, Chair, Division of Pulmonary and Critical Care Medicine; Associate Chair, Department of Medicine, University of Maryland, Baltimore
Other Study IDs: HP-00110218
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Lung Cancer Screening; Healthy Volunteers (HV); Unhealthy Volunteers
Keywords: Lung Cancer; Lung Cancer Screening; Healthy Volunteers; Unhealthy Volunteers
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Study Population 1: This study population will consist of individuals who have a new diagnosis of lung cancer and have not received chemotherapy treatment for their lung cancer. Individuals who have received surgical resection or stereotactic body radiation therapy (SBRT) for their lung cancer will be included.
  Interventions: Other: Epigenetic Signature Assay
- Study Population 2: This study population will consist of individuals who have a diagnosis of lung cancer and have received chemotherapy treatment for their lung cancer. All stages of lung cancer will be included including individuals in remission.
  Interventions: Other: Epigenetic Signature Assay
- Study Population 3: This study population will consist of individuals who are at high risk of developing lung cancer, such as people with a long smoking history, and are receiving yearly lung screening scans.
  Interventions: Other: Epigenetic Signature Assay
- Study Population 4: This study population will consist of individuals who may be hospitalized for another condition such as pneumonia or heart failure at time of enrollment into the study. Individuals who have a greater than 10 pack year history of smoking will not be included in this population.
  Interventions: Other: Epigenetic Signature Assay
- Study Population 5: This study population will consist of individuals who have no other significant medical problems.
  Interventions: Other: Epigenetic Signature Assay

INTERVENTIONS:
Other: Epigenetic Signature Assay — Up to 15 ml of blood will be collected from each patient at various time points throughout their 5 years of participation. DNA extraction, bisulfite conversion and analysis of epigenetic markers through PCR or next-generation sequencing will be performed. An epigenetic signature assay will then be identified.

SUMMARY:
The purpose of this research study is to test a new process for diagnosing lung cancer by examining changes to your DNA that can be detected from a blood test. The information we learn by doing this study could potentially help people in the future.

Participants in this study will have blood samples collected, have their medical records reviewed by study personnel and fill out questionnaires at different time points during the study. Blood sample collection will occur during normal routine clinic visits. Participation in this study will last approximately 5 years.

DETAILED DESCRIPTION:
This clinical testing research study outlines the validation process for an epigenetic assay targeting host peripheral blood cell and the associated host DNA methylation signatures designed to diagnose lung cancer. The overall protocol process will involve three distinct stages representing three patient cohorts with up to 250 subjects per cohort across 5 populations of patients. Cohort one will act as signature development phase; cohort two will act as signature finalization phase; and cohort three will act as a validation cohort phase. Each cohort will include the following patient populations with up to 50 patients per population:

1. Lung cancer; No chemotherapy. Surgical resection or stereotactic body radiation therapy (SBRT) only
2. Lung cancer; With chemotherapy. All stages including remission
3. At risk group (Lung cancer screening population)
4. Control group with mixed comorbid disease EXCLUDING tobacco use of greater than 10 pack years (PY) or chronic obstructive pulmonary disease (COPD)
5. Healthy controls with no comorbid disease

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Patient at University of Maryland Baltimore Washington Medical Center
* Willing and able to consent to study procedures listed in the protocol
* Ability to speak and understand English

Exclusion Criteria:

* Younger than 18 years old
* Patient not cared for at University of Maryland Baltimore Washington Medical Center
* Unable to consent to study procedures listed in the protocol
* Unable to speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from patients being cared for at the University of Maryland Baltimore Washington Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Identification of tumor-associated host methylation signature | 5 years
  Genome-wide methylation profile of whole blood from lung cancer patients, pre-cancer patients, patients undergoing therapy, and control subjects.
Technology development | 5 years
  The investigators will develop array-based assays using whole-blood samples, focused on disease-specific methylation sites to provide early diagnosis, prognosis, and therapeutic efficacy prediction.
Technology validation | 1 year
  The investigators will validate identified blood-based circulating methylation signatures in patients with undiagnosed pulmonary nodules.

SECONDARY OUTCOMES:
EORTC QLQ-C30 Questionnaire | 5 years
  The European Organization for Research and Treatment of Cancer core quality of life questionnaire, (EORTC QLQ-C30) is a cancer-specific quality of life instrument designed to assess health-related quality of life of cancer patients and is intended to be supplemented by disease-specific questionnaires, such as the lung cancer specific module, the EORTC QLQ-LC13. The EORTC QLQ-C30 incorporates nine multi-item scales including five functional scales (Physical, Role, Cognitive, Emotional and Social Functioning); three symptom scales (Fatigue, Pain and Nausea/Vomiting); and a Global Health Status/QoL scale. Six single item scales are also included (Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea and Financial Difficulties). All of the scales and single-item measures range in score from 0 to 100. A higher score represents a higher level of symptom burden.
EORTC QLQ-LC13 Questionnaire | 5 years
  The European Organization for Research and Treatment of Cancer quality of life questionnaire module on Lung Cancer, EORTC QLQ-LC13, is a supplementary questionnaire meant to be used in conjunction with the full QLQ-C30. The QLQ-LC13 incorporates one multi-item scale to assess dyspnea, and a series of single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All of the scales and single-item measures range in score from 0 to 100. A higher score represents a higher level of symptom burden.
SF-36v2 Questionnaire | 5 years
  The short-form of 36 questions (SF-36v2) is a multipurpose, 36-item survey that measures eight domains of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It yields scale scores for each of these eight health domains, and two summary measures of physical and mental health. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore Washington Medical Center, Glen Burnie, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Fan Z, Meng Y, Liu S, Zhan H. Blood-based DNA methylation signatures in cancer: A systematic review. Biochim Biophys Acta Mol Basis Dis. 2023 Jan 1;1869(1):166583. doi: 10.1016/j.bbadis.2022.166583. Epub 2022 Oct 18. PMID 36270476
- [Background] Terp SK, Stoico MP, Dybkaer K, Pedersen IS. Early diagnosis of ovarian cancer based on methylation profiles in peripheral blood cell-free DNA: a systematic review. Clin Epigenetics. 2023 Feb 14;15(1):24. doi: 10.1186/s13148-023-01440-w. PMID 36788585
- [Background] Ibrahim J, Peeters M, Van Camp G, Op de Beeck K. Methylation biomarkers for early cancer detection and diagnosis: Current and future perspectives. Eur J Cancer. 2023 Jan;178:91-113. doi: 10.1016/j.ejca.2022.10.015. Epub 2022 Oct 27. PMID 36427394
- [Background] Guo Y, Yin J, Dai Y, Guan Y, Chen P, Chen Y, Huang C, Lu YJ, Zhang L, Song D. A Novel CpG Methylation Risk Indicator for Predicting Prognosis in Bladder Cancer. Front Cell Dev Biol. 2021 Sep 1;9:642650. doi: 10.3389/fcell.2021.642650. eCollection 2021. PMID 34540821
- [Background] Xie Y, Li P, Sun D, Qi Q, Ma S, Zhao Y, Zhang S, Wang T, Wang J, Li S, Gong T, Xu H, Xiong M, Li G, You C, Luo Z, Li J, Wang C, Du L. DNA Methylation-Based Testing in Peripheral Blood Mononuclear Cells Enables Accurate and Early Detection of Colorectal Cancer. Cancer Res. 2023 Nov 1;83(21):3636-3649. doi: 10.1158/0008-5472.CAN-22-3402. PMID 37602818
- [Background] Wang T, Li P, Qi Q, Zhang S, Xie Y, Wang J, Liu S, Ma S, Li S, Gong T, Xu H, Xiong M, Li G, You C, Luo Z, Li J, Du L, Wang C. A multiplex blood-based assay targeting DNA methylation in PBMCs enables early detection of breast cancer. Nat Commun. 2023 Aug 7;14(1):4724. doi: 10.1038/s41467-023-40389-5. PMID 37550304